CLINICAL TRIAL: NCT00684879
Title: Illness Perceptions and the Health Belief Model: Screening Behavior in Adults With Hereditary Hemorrhagic Telangiectasia
Brief Title: Screening Behavior in Adults With Hereditary Hemorrhagic Telangiectasia
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908143; 08-HG-N143
Record Dates: First submitted 2008-05-24; First posted 2008-05-28 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2016-01-07

CONDITIONS: Osler-Rendu-Weber Disease; Osler-Rendu Disease; Telangiectasia, Hereditary Hemorrhagic
Keywords: Hereditary Hemorrhagic Telangiectasia; Health Belief Model; Illness Perceptions; Screening; HHT
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will explore the factors that influence screening behaviors of adults diagnosed with hereditary hemorrhagic telangiectasia (HHT), an inherited condition in which blood vessel defects called arteriovenous malformations (AVMs) result in direct connections between arteries and veins. Patients most commonly have small AVMs called telangiectases on the tongue, face, hands, mouth, and throat and the mucosal linings of the nose and gastrointestinal tract. Recurrent nosebleeds are a hallmark of the disease. Large AVMs can also occur in various organs, causing sudden and life-threatening complications.

The study will examine how patients think and feel about their condition and what actions they take to screen for internal symptoms of the disease.

Men and women 18 years of age and older who have HHT may be eligible for this study. Participants fill out a 30-minute questionnaire, available in print or online, that includes questions about the participant s

* beliefs about HHT
* actions taken to screen for internal symptoms of HHT
* experience with HHT
* current health status, family history and demographic information

DETAILED DESCRIPTION:
The proposed study aims to understand the factors that influence screening behaviors of adults with hereditary hemorrhagic telangiectasia (HHT). HHT is a chronic condition, but with early diagnosis followed by adherence to recommended screening guidelines, the major complications of this disorder can be avoided and disability or even death can be prevented. Yet, it has come to the attention of healthcare professionals that the recommended screening is not commonly followed by individuals with HHT, even when the risk of serious complications is known. Nonadherence to screening recommendations is not unique to HHT. It is rather common across chronic conditions, and genetic diseases, such as HHT, are no exception. However, HHT may have an added barrier to screening and treatment adherence in that it is a rare and underdiagnosed condition. Inadequate knowledge of healthcare providers may be a serious barrier to prevention, diagnosis, and treatment. The Health Belief Model (HBM) can be used to frame this study of HHT screening. The HBM posits that preventive health behaviors will be acted upon if individuals regard themselves as susceptible to the threat, they believe the consequences to be severe, and the perceived benefits outweigh the perceived barriers. In addition to the HBM constructs, this study will also consider the role of illness representations which provide a more personal view of the lived experience of individuals with HHT. A cosss-sectional design will be used to investigate the relationships among the domains of illness representations, HBM constructs (perceived susceptibility, perceived benefits, barriers, self-efficacy, response efficacy, cues to action), and HHT-specific screening guidelines. Participants will be recruited from the HHT Foundation International, Inc., an outline HHT Awareness social group, and HHT Clinics. Participants will be asked to complete either a web-based or a paper survey. The main outcome measure is screening behaviors and intentions to screen for complications associated with HHT.

ELIGIBILITY:
* INCLUSION CRITERIA:

Men and women who self-report having a diagnosis of HHT.

To read and write English.

EXCLUSION CRITERIA:

Individuals younger than 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2008-05-21; Study Completion 2016-01-07

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bayrak-Toydemir P, Mao R, Lewin S, McDonald J. Hereditary hemorrhagic telangiectasia: an overview of diagnosis and management in the molecular era for clinicians. Genet Med. 2004 Jul-Aug;6(4):175-91. doi: 10.1097/01.gim.0000132689.25644.7c. PMID 15266205
- [Background] Guttmacher AE, Marchuk DA, White RI Jr. Hereditary hemorrhagic telangiectasia. N Engl J Med. 1995 Oct 5;333(14):918-24. doi: 10.1056/NEJM199510053331407. No abstract available. PMID 7666879
- [Background] Rand CS. Measuring adherence with therapy for chronic diseases: implications for the treatment of heterozygous familial hypercholesterolemia. Am J Cardiol. 1993 Sep 30;72(10):68D-74D. doi: 10.1016/0002-9149(93)90014-4. PMID 8213501